CLINICAL TRIAL: NCT01048814
Title: Retrospective Study to Develop a Training Set for a Cross Validated Chemoresponse Marker Algorithm in Cases With Ovarian, Peritoneal or Fallopian Tube Cancer
Brief Title: Retrospective Case Study to Validate Existing Chemoresponse Marker Test in Ovarian, Peritoneal or Fallopian Cancer Cases
Status: Completed | Type: Observational
Sponsor: Precision Therapeutics (Industry)
Responsible Party: Holly Gallion, MD, Precision Therapeutics
Other Study IDs: PT-103
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian, Peritoneal, Fallopian Cancer: Recurrent, Peristent or Refractory
  Interventions: Other: ChemoFx

INTERVENTIONS:
Other: ChemoFx — Chemoresponse Marker Assay

SUMMARY:
The purpose of this study is to improve upon and validate the prognostic and/or predictive accuracy of a drug response marker by the development of improved alternative algorithms based on the actual clinical outcome of retrospective cases.

DETAILED DESCRIPTION:
This is a multicenter, retrospective chart review study of de-identified drug response marker results and a limited data set of clinical outcome data. Data from approximately 512 cases will be collected from approximately 30 sites and correlated to the secondary endpoints identified in order to produce a training set that will incorporate additional improvements to the existing ChemoFx scoring system. The outcome of progression free survival will be defined as the period of time between the first dose of chemotherapy following the report of the marker result until clinical progression or death. Objective response will be measured from the first dose of chemotherapy following the report of the marker result until progression or change in therapy.

ELIGIBILITY:
Inclusion Criteria:

* Case has an original pathology report showing, epithelial ovarian, peritoneal, or fallopian tube carcinoma.
* Cases must meet one of the following classifications: Recurrent: Complete Response following primary therapy and a period of absence of no measurable disease; Persistent: Partial Response following 6 cycles of a platinum based therapy with measurable disease remaining or Refractory: Stable Disease or Progressive Disease during primary platinum therapy.
* Case must have a commercial ChemoFx drug response marker final report

Exclusion Criteria:

* Cases with evidence of synchronous primary endometrial cancer or a past history of primary endometrial cancer are excluded unless all of the following conditions are met: Stage not greater than I-B; Less than 3 mm invasion without vascular or lymphatic invasion; No poorly differentiated subtype, including papillary serous, clear cell, or other FIGO Grade 3 lesion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 512 cases of ovarian, peritoneal or fallopian tube, recurrent, persistent, or refractory cancer that have had ChemoFx drug response marker results for NCCN recommended second line therapy from August 2006 to January 31, 2009 will be included in the compilation of the training set. Cases will be selected sequentially from each participating clinical site.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Gallion, MD, Study Director — Vice President, Clinical Affairs
Locations (1):
- Precision Therapeutics, Inc., Pittsburgh, Pennsylvania, United States